CLINICAL TRIAL: NCT01075958
Title: The Relationship Between Serum PUFAs and Cognitive Function in Healthy Young Adults
Brief Title: Polyunsaturated Fatty Acids (PUFA) Status and Cognitive Function in Healthy Young Adults
Status: Completed | Type: Observational
Sponsor: Northumbria University (Other)
Responsible Party: Philippa Jackson, Northumbria University
Other Study IDs: 16N3
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Attention; Memory; Mood; Mental Fatigue
Keywords: n-3 PUFAs; Fish oil; Cognitive function; Healthy young adults
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
To date, the relationship between omega-3 polyunsaturated fatty acids (n-3 PUFAs) in cognitively intact individuals has only been examined in a limited number of studies; it is at present unknown whether supplementation with n-3 PUFAs can improve cognitive function and mood in this population. Further to this, it still remains to be established whether a relationship exists between peripheral fatty acid status-reflective of dietary n-3 PUFA intake-and cognitive function in this population. The current study therefore aims to address this issue by exploring the relationship between serum PUFAs and specific cognitive functions in a sample of healthy adults. To this end, participants will complete a range of cognitive tasks evaluating performance across the domains of attention, memory and executive function. Self-report mood assessments will be included as secondary measures.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* 18-35 years
* Healthy
* No herbal supplements/prescription medications (excl. contraceptive pill)
* Non smoker
* Native English speaker

Exclusion Criteria:

* BMI ≥ 30

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample will be drawn from a student and professional population in the Newcastle upon Tyne area in the UK
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa A Jackson, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- See also: Brain, Performance and Nutrition Research Centre, Northumbria University — http://www.nutrition-neuroscience.co.uk/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place on the Northumbria University campus via posted adverts and email messages sent using the university distribution lists. Recruitment took place in 2 waves; the first taking place between July 31 - November 8 2007, and the second between March 26 - September 9 2008.
Pre-assignment Details: Participants from whom a venous blood sample could not be obtained were not entered into the analysis.
Groups:
- Healthy Participants: Participants declared themselves as healthy, a non-smoker and prescription and herbal medication free.
Period: Overall Study
Arm/Group | Healthy Participants
Started | 283
Completed | 239
Not Completed | 44
Not completed — Blood sample could not be obtained | 44

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Participants
Number analyzed (Participants) | 283
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 283
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 22.47 (3.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187
  Male | 96
Region of Enrollment [Number; unit: participants]
  United Kingdom | 283

OUTCOME MEASURES:

1. Primary Outcome: Simple Reaction Time (Attention)
Description: The participant was instructed to press the 'space bar' on the laptop keyboard as quickly as possible every time an upwards pointing arrow appeared on screen. Fifty stimuli were presented with an inter-stimulus duration that varied randomly between 1 and 3.5 seconds.
Time Frame: Single visit
Population: Only those participants for whom a venous blood sample was obtained (N=239) were entered into the analysis. A further 20 participants were excluded on the basis that their BMI exceeded 30, and could not be considered 'healthy individuals'.
Measure: Mean (Standard Error); unit: ms
Groups:
- Healthy Participants: All eligible participants.
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
ms | 287.7 (2.67)

2. Secondary Outcome: Depression, Anxiety and Stress Scale (DASS)
Description: The DASS is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress. Each of the three DASS scales contains 14 items. Subjects are asked to use 4-point (0-3) severity/frequency scales to rate the extent to which they have experienced each state over the past week. Scores for Depression, Anxiety and Stress (0-42) are calculated by summing the scores for the relevant items, with higher scores indicating higher incidence of negative emotional symptoms. A total score can be derived by adding scores from each of the subscales (0-126).
Time Frame: Single visit-90 minutes
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
Scores on a scale | 22.45 (16.70)

3. Primary Outcome: Choice Reaction Time (Attention)
Description: An arrow appeared on the screen pointing to the left or to the right. Participants responded with a left or right key press corresponding to the direction of the arrow. There was a randomly varying inter-stimulus interval of between 1 and 3 seconds for a total of fifty stimuli.
Time Frame: Single visit
Measure: Mean (Standard Error); unit: ms
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
ms | 412.79 (3.75)

4. Primary Outcome: Four Choice Reaction Time (Attention)
Description: A visual representation of the four direction arrow keys of a standard keyboard was presented on screen. The arrows 'lit up' at random on screen until the corresponding key press was made. In all, each arrow was the target stimulus 12 times, forming a total of 48 stimuli for this task in all.
Time Frame: Single visit
Measure: Mean (Standard Error); unit: ms
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
ms | 499.52 (5.84)

5. Primary Outcome: Numeric Working Memory (Working Memory)
Time Frame: Single visit
Measure: Mean (Standard Error); unit: percent of correct responses
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
percent of correct responses | 95.57 (0.34)

6. Primary Outcome: Alphabetic Working Memory (Working Memory)
Description: Five random letters (A-Z) were presented sequentially for the participant to hold in memory. This was followed by a series of 30 probe digits (15 targets and 15 distractors) for each of which the participant indicated whether or not it had been in the original series by a simple key press. The task consisted of 3 separate trials.
Time Frame: Single visit
Measure: Mean (Standard Error); unit: percent of correct responses
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
percent of correct responses | 94.5 (0.30)

7. Primary Outcome: Corsi Blocks Span (Spatial Working Memory)
Description: In this task nine identical blue squares appeared on screen in non-overlapping random positions. A set number of blocks changed colour from blue to red in a randomly generated sequence. Participants were instructed to repeat the sequence by clicking on the blocks using the mouse and cursor. The task was repeated five times at each level of difficulty. The sequence span increased from 4, until the participant could no longer correctly recall the sequence, resulting in a span measure of nonverbal working memory, calculated by averaging the level of the last five correctly completed trials.
Time Frame: Single visit
Measure: Mean (Standard Error); unit: Blocks remembered in sequence
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
Blocks remembered in sequence | 5.90 (0.08)

8. Primary Outcome: 3-back Task (Working Memory)
Description: A continuous string of letters (upper and lower case; inter-stimulus interval of 2.5 seconds) was presented; 45 letters in total with 15 target pairs. For each stimulus, participants were instructed to indicate whether this was the same letter that appeared three letters before.
Time Frame: Single visit
Measure: Mean (Standard Error); unit: percent of correct responses
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
percent of correct responses | 80.89 (1.04)

9. Primary Outcome: Immediate Word Recall (Episodic Memory)
Description: A unique set of fifteen words is presented. Words were selected at random from a large bank of words derived from the MRC Psycholinguistic Database matched for word length, frequency, familiarity and concreteness. Stimulus duration was one second, as was the inter-stimulus duration. Following word presentation, the participant was allowed 60 seconds to write down as many of the words as possible.
Time Frame: Single visit
Measure: Mean (Standard Error); unit: Number of words recalled
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
Number of words recalled | 6.21 (0.16)

10. Primary Outcome: Delayed Word Recall (Episodic Memory)
Description: The participant was again given 60 seconds to write down as many of the words presented previously as possible.
Time Frame: Single visit
Measure: Mean (Standard Error); unit: Number of words recalled
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
Number of words recalled | 4.73 (0.16)

11. Primary Outcome: Word Recognition (Episodic Memory)
Description: The original 15 words plus 15 distractor words were presented one at a time in a random order. For each word the participant indicated whether or not it was included in the original list of words by pressing appropriate 'yes' and 'no' keys as quickly as possible. Stimuli remained on screen until an appropriate response had been made.
Time Frame: Single visit
Measure: Mean (Standard Error); unit: percent of correct responses
Arm/Group | Healthy Participants
Number analyzed (Participants) | 219
percent of correct responses | 80.35 (0.68)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected only on the day of testing.
Description: The testing day comprised a single 90 minute session.
Arm/Group | Healthy Participants
Serious Adverse Events (participants affected / at risk) | 0/283
Other Adverse Events (participants affected / at risk) | 0/283

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No